CLINICAL TRIAL: NCT00936117
Title: Phase II Study of the Pharmacokinetics of Posaconazole Prophylaxis in Relapsed or Refractory Patients With Acute Leukemia
Brief Title: Pharmacokinetics of Posaconazole Prophylaxis in Acute Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0793
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Leukemia; Fungal Infection
Keywords: Cancer of the Blood; Cancer of Bone Marrow; Acute Leukemia; AML; Fungal infection; Prophylaxis; Posaconazole; SCH 56592; Noxafil; Chemotherapy
MeSH Terms: conditions — Leukemia; Mycoses; Bone Marrow Neoplasms | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Posaconazole (Experimental): Posaconazole 200 mg (liquid) by mouth 3 times per day.
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — 200 mg (liquid) by mouth 3 times per day.
  Other Names: SCH 56592; Noxafil

SUMMARY:
The goal of this clinical research study is to learn the amount of posaconazole that is in the body at different time points when given to patients with leukemia. The safety of this drug will also be studied.

Objectives:

Primary:

To study the plasma pharmacokinetics of posaconazole in patients with newly diagnosed acute myelogenous leukemia (AML) or high-risk myelodysplastic syndrome (HR-MDS) undergoing induction chemotherapy or relapsed or refractory patients who will receive salvage chemotherapy.

Secondary:

To evaluate the safety of posaconazole given as prophylaxis.

DETAILED DESCRIPTION:
Chemotherapy can lower immune system function, which can cause fungal infections to occur more easily. The standard treatment for prevention of such infections includes drugs such as voriconazole and liposomal amphotericin B that help prevent fungus from growing.

The Study Drug:

Posaconazole is designed to block the ergosterol synthesis (a part of the fungal membrane). This may help to prevent fungal infections.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take posaconazole by mouth 3 times per day. Posaconazole is a liquid. You should take the study drug after a full meal or with a liquid nutritional supplement (such as a protein shake). If you are not able to eat food, you should take it with a carbonated beverage (such as soda).

Food and Drug Diary:

You will be also be given a food and drug diary where you will write down the time you took each dose. You should also record the time eaten and describe what you ate or drank at each meal. This information will be used to find out the number of calories and amount of protein, carbohydrates, and fat you have consumed. You will be given a small bag where you can keep the drug and diary. You should return this diary after the last blood draw.

Blood Draws for Pharmacokinetics (PK) Testing:

While you are on study, blood (about 1 teaspoon each time) will be drawn for PK testing. PK testing measures the amount of study drug in the body at different time points.

* Days 1, 3, and 10, before your first dose of study drug and 3, 5, and 10 hours after the first dose of the day
* Days 2 and 4, about 24 hours after the first dose the day before

Blood (about 1 teaspoon) will also be drawn for PK testing 1 time at any of the following time points:

* Before you start a new dose of study drug, if the dose needs to be raised
* If you stop taking the study drug due to intolerable side effects or a fungal infection

Note that if you are not already in the hospital on the days of the PK blood draws, you will need to stay at the hospital for about 10 hours on these days.

Length of the Study:

You will take the study drug for up to 42 days. You will be taken off study if you experience intolerable side effects, if you develop an invasive fungal infection, or if the doctor thinks it is in your best interest.

This is an investigational study. Posaconazole is FDA approved and commercially available for the prevention of fungal infections.

Up to 25 patients will take part in the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients newly diagnosed with AML or high-risk MDS undergoing induction chemotherapy or refractory or relapsed patients with AML or high-risk MDS who will receive first or second salvage chemotherapy. (Salvage patients are defined as patients that achieved remission and relapsed or patients who were refractory to initial frontline chemotherapy)
2. Age > 18 years and able to take oral intake.
3. Patients must sign an informed consent.
4. Patients agree to medically approved forms of contraception
5. Patients on prior antifungal prophylaxis with voriconazole, itraconazole or fluconazole are eligible if they completed 3 days wash-out period if on voriconazole, or 14 days wash-out period if on itraconazole or 7 days wash-out period if on fluconazole

Exclusion Criteria:

1. Patients with history of anaphylaxis attributed to azole compounds
2. Patients with clinical or other evidence that indicates that they have proven or probable invasive fungal infection prior to enrollment (EORTC criteria)
3. Patients with baseline total bilirubin levels > 3 times the upper normal limits (i.e. > 3.0 mg/dl); or baseline SGPT > 5 times upper limit normal.
4. Patients receiving any medication that is contraindicated with the use of posaconazole
5. Patients with baseline creatinine levels NCI grade 3 or above (> 3.0 - 6.0 X ULN)
6. Patients with baseline QTc prolongation NCI grade 1 or above (QTc > 0.45 - 0.47 seconds).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 30, 2009 to January 3, 2011. From January 2010 through August 2010, adult with newly diagnosed acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (HR-MDS) undergoing induction chemotherapy or first salvage therapy were recruited at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 25 participants enrolled, five participants were excluded from the trial -- two were ineligible, one withdrew consent before start of treatment, another two were excluded from the study for other reasons.
Period: Overall Study
Arm/Group | Posaconazole
Started | 20
Completed | 10 (Completed 42 days on study drug)
Not Completed | 10
Not completed — Adverse Event | 7
Not completed — Unable to continue oral medication | 3

BASELINE CHARACTERISTICS:
Arm/Group | Posaconazole
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 65 [34 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20
Participant Diagnosis [Number; unit: participants]
  AML, Induction | 19
  AML, Relapse | 1
Chemotherapy Received [Number; unit: participants] — Participant's first induction chemotherapy, either with a clofarabine-based regimen or a cytarabine-based regimen. Exception listed as miscellaneous chemotherapy treatment, and include AZD1152 (an experimental aurora kinase inhibitor) alone (1 participant) or in combination with low-dose cytarabine (2 participants).
  participants
    Cytarabine-containing regimen | 9
    Clofarabine-containing regimen | 8
    Miscellaneous* | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration in Plasma (Cmax)
Description: Pharmacokinetic samples were obtained on day 1, day 3 and day 10 of prophylaxis. A total of 15 samples (3 ml each sample) per participant were obtained, with thrice daily dosing planned around standard meal times. On day 1 and day 3 of prophylaxis sampling was done pre dose (0), and at 3, 5, 10 and 24 hours (±10 minutes) post dose from the time of the first dose of the day. On day 10 of prophylaxis sampling was done pre dose (0), and at 3, 5, and 10 hours (±10 minutes) post dose from the time of the first dose of the day.
  Posaconazole levels were assayed by high performance liquid chromatography (HPLC). The testing range for posaconazole is from 125 - 5000 ng/ml. There are no established therapeutic ranges for posaconazole.
Time Frame: Pharmacokinetics: Day 1, Day 3 and Day 10 of prophylaxis.
Population: Of the 11 females enrolled, one was not evaluable for the outcome thus excluded from analysis.
Measure: Median (Full Range); unit: ng/ml
Groups:
- Posaconazole (Females); Posaconazole (Males): Posaconazole 200 mg (liquid) by mouth 3 times per day.
Arm/Group | Posaconazole (Females) | Posaconazole (Males)
Number analyzed (Participants) | 10 | 9
ng/ml
  Day 2, Hour 24 | 200 [140 to 660] | 290 [120 to 770]
  Day 4, Hour 24 | 300 [140 to 1820] | 580 [260 to 1090]
  Day 9, Hour 24 | 770 [140 to 2450] | 800 [370 to 1690]

ADVERSE EVENTS:
Time Frame: Adverse event data collected to 42 days following start of treatment, overall study period January 19, 2010 to February 11, 2011.
Description: The adverse events presented below reflect all SAEs and AEs reported by participants, regardless of whether events were treatment-related or non-treatment-related.
Arm/Group | Posaconazole
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=20)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Acid Reflux (Gastrointestinal disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurry Vision (Eye disorders) | 1 (1)
Body Aches (General disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Dysuria (Renal and urinary disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Elevated Alanine Aminotransferase (ALT) (Metabolism and nutrition disorders) | 1 (1)
Elevated Bilirubin (Metabolism and nutrition disorders) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Fungal Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Intracranial Hemmorrhage (Nervous system disorders) | 1 (1)
Mouth Sores (Gastrointestinal disorders) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Nausea/Vomiting (Gastrointestinal disorders) | 8 (9)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Testicular Cyst (Reproductive system and breast disorders) | 1 (1)
Transaminitis (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes